CLINICAL TRIAL: NCT06269952
Title: Intimate Partner Violence Among People Who Inject Drugs - Prevalence, Risk Factors and Experiences
Status: Recruiting | Type: Observational
Sponsor: Region Stockholm (Other Government)
Responsible Party: Sponsor
Other Study IDs: MVarmafalk
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Intimate Partner Violence (IPV); People Who Inject Drugs
Keywords: intimate partner violence; domestic violence; people who inject drugs

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People who inject drugs: People who inject drugs, over 18 years of age, that participate in the needle syringe program in Stockholm, Sweden
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention. The participants are asked questions from and questionnaire and later also interviewed guide by an interview-guide

SUMMARY:
There are around 15,6 million people who inject drugs (PWID) worldwide, of which around 3,5 million are women who inject drugs (WWID) (1). In Sweden, estimates suggest 8000-21000 PWID (2). PWID are exposed to substantial health risks that are directly linked to injection drug use, such as blood borne viruses (hepatitis and HIV), overdoses and skin and tissue infections. Additionally psychiatric disorders are common and PWID's general health is often neglected (3,4,5).

In Sweden, harm reduction units such as needle and syringe programs (NSP) have scaled-up in recent years. In Stockholm the first NSP opened in 2013 and the second in 2018. In 2022, 4600 individuals were enrolled in the program since it opened, of which approximately 25% were women. Around 2000 were active participants, defined as having visited the program at least once during the last 12 months. In 2021 54% of the participants stated amphetamine as the last drug injected, 31% heroin, 4% buprenorphine and 11% other drugs. Most participants were between 30-49 years of age. In addition to distribution of sterile needles and injection paraphernalia, the NSP staff (nurses, doctors, midwifes, counselors) provides services such as testing for blood borne viruses, vaccinations, wound care, take-home naloxone, reproductive health services, counselling, support in contact with social service and referrals for substance use disorder treatment and hepatitis C/HIV treatment.

Gender-based violence (GBV) is a global health issue and WHO estimates that one in three women globally have been exposed to some sort of partner violence during their lifespan (7). Intimate partner violence (IPV) is defined as violent behavior between two people who have a close relationship, such as partners, ex-partners, siblings, relatives, friends and alike. In Sweden around 14% of women and 5% of men are exposed to physical violence in an intimate partner relationship during their lifespan however 20-25% of women and around 17% of men are exposed to psychological violence during their lifespan (8; 9). The prevalence of IPV among PWID is estimated to be significantly higher than in the general population (10). A study from USA found the risk of IPV to be three times higher and the prevalence estimated between 35-57% (7). In international studies, IPV exposure is found to be a significant risk factor for needle sharing among WWID (11, 12). There are other well-known consequences of IPV including impact on sexual and reproductive health rights, physical and psychological wellbeing, increased risk of contracting HIV and hepatitis C (13; 14). IPV exposure disproportionately affects WWID worldwide, however studies in Sweden on IPV exposure in the PWID population is scarce. To date there are studies that address this among women with substance use disorders but none with an exclusive focus on PWID or WWID. In clinical research of women diagnosed with substance use disorders (SUD) with psychiatric comorbidities and social challenges, one study indicates that the majority (91%, n=79) of women had been exposed to some form of IPV (15). Another study of women with SUD (n=52), 50% reported exposure of serious violence and the majority (96%) reported exposure to psychological violence (10). There are different types of IPV; psychological, physical, sexual, financial, latent, digital, neglect, honor related, aftermath of IPV (16). Our research team has previously carried out a qualitative interview study among WWID at the Stockholm NSP in 2019 to investigate reasons and barriers for participation among women (17). The interviews illustrated that IPV is common. In the proposed studies, for this doctoral thesis, we have chosen to focus on physical, sexual, psychological and financial violence among PWID motivated by findings in our previous research.

PWID and specifically WWID are regarded as groups who are especially vulnerable for IPV exposure and should therefore be prioritized in the national efforts to prevent IPV (15). However, there are no studies estimating the prevalence and frequency of IPV among PWID in Sweden. Previous international studies suggest that PWID are exposed to IPV to a greater extent than the general population, and women with substance use disorders are exposed to an alarming degree of violence (15). In Sweden there are no tailored interventions for PWID or WWID who are exposed to IPV, it is reasonable to believe that there is a need for a multi-faceted program for PWID exposed to IPV, however this is still unexplored.

The overall aim of this project is to increase knowledge about IPV among PWID and WWID as particularly vulnerable groups in regards to IPV. More specifically, the aim is to investigate the prevalence and frequency of different types of IPV among PWID at the Stockholm NSP and to explore the experiences' of IPV, needs and preferences for IPV support among WWID to facilitate tailored support and prevention programs for those exposed.

ELIGIBILITY:
Inclusion Criteria: at least 18 years of age, injecting drugs, participating in the needle syringe program in Sweden

-

Exclusion Criteria:

* under the age of 18
* heavily intoxicated
* psychotic symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who inject drugs, both male and female, and other (non-binary, not-known) participating in the needle syringe program in Stockholm, Sweden. Interviews with women and non-binary people specifically, as an extra vulnerable group
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-10-05 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants exposed to physical intimate partner violence | 1 year
  A questionnaire will be used to collect data on exposure to different types of intimate partner violence. In this case physical intimate partner violence
Number of participants exposed to psychological intimate partner violence | 1 year
  A questionnaire will be used to collect data on exposure to psychological intimate partner violence, during the last 12 months and the participants whole lifespan.
Number of participants exposed to sexual intimate partner violence | 1 year
  A questionnaire will be used to collect data on exposure to sexual intimate partner violence, during the last 12 months and the participants whole lifespan.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Strömdahl, M.D, Associate Professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Needle syringe program, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No